CLINICAL TRIAL: NCT03354897
Title: Clinical Study of UMOD NKCC2 Interaction on Salt-sensitivity in Hypertension
Acronym: UMOD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN14CE400
Record Dates: First submitted 2017-09-28; First posted 2017-11-28 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Diseases; Hypertension
Keywords: stratified medicine, UMOD, torasemide
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — Torsemide; Tablets

STUDY DESIGN:
Intervention Model Description: This study is a multi-centre prospective cohort study to investigate whether individuals possessing the AA genotype of the single nucleotide polymorphism, rs13333226, are better responders to loop diuretics compared to those possessing the G allele.
Masking Description: prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): 16 weeks treatment 5mg/day
  Interventions: Drug: Torasemide 5Mg Tablet

INTERVENTIONS:
Drug: Torasemide 5Mg Tablet — 16 weeks treatment

SUMMARY:
The hypothesis is based on UMOD rs13333226 genotype, there are two strata of hypertensive patients. The High-UMOD group (AA genotype) has increased UMOD excretion, greater salt sensitivity, HTN, normal eGFR and greater BP response to loop diuretics like furosemide. The Low-UMOD group (G allele) has decreased UMOD excretion, salt resistance, increased eGFR, increased proximal tubular reabsorption of Na (possibly related to increased GFR), a poor BP response to loop diuretics, and possibly diminished function of NKCC2. The High-UMOD strata will have decreased delivery of Na+ to the distal tubule and collecting duct because NKCC2 function is normal and the study hypothesis is that the participants will be more responsive to loop diuretics. In contrast, the Low-UMOD group (G allele) will not show a similar response to loop diuretics. This may be related either to lower Na delivery to the TAL, because of increased proximal tubular reabsorption of Na+, or a suppressed function of NKCC2. The population distribution of the High-UMOD group (AA) is 67%. Our overall objective is to test the hypothesis that hypertensive subjects with uncontrolled HTN open possessing the AA genotype of rs13333226 will be better responders to loop diuretics compared to those possessing the G allele.

DETAILED DESCRIPTION:
There are over 1 billion people with HTN worldwide, and the World Health Organisation suggests this will rise to 1.5 billion by 2020.(1) Up to 30% of hypertensive patients have resistant HTN (uncontrolled BP on > 3 drugs of which one must be a diuretic) and ~50% have uncontrolled HTN, with a 7-fold higher cardiovascular risk.

In clinical practice, criteria such as ancestry and serum renin levels provide only a rough indication of the underlying disease pathway and, while pharmacotherapy is the mainstay of HTN management, the selection of antihypertensive therapy is essentially by trial-and-error. Five drug classes are the main first-line agents for HTN, but response rates to any given drug are only ~50%. There are no new anti-hypertensive drugs in clinical trials and there is a need to either develop newer agents or target existing drugs to specific strata of hypertensive patients in whom they would be beneficial. The recent failure of the Renal Sympathetic Denervation trial, which used a novel device strategy for resistant HTN, highlights the limited options available in the management of uncontrolled or resistant HTN.

HTN as a phenotype demonstrates stratification in the population, based on the specific pathophysiological and molecular pathways that are operative and this is reflected in the current NICE guidelines. However, there has been little progress in stratification by leveraging genomic and molecular information, although there is evidence that this may be useful. Monogenic forms of HTN show that identification of the many causative mutations, primarily affecting the kidney and sodium balance, can inform therapy - for example, glucocorticoids in glucocorticoid remediable aldosteronism and amiloride in Liddle syndrome. Despite the successful adoption of the BHS/NICE treatment algorithm for the treatment of HTN, there remains substantial clinical uncertainty about the preferred clinical management of people with uncontrolled or treatment resistant HTN. Moreover, the choice of diuretic, suggested in HTN guidelines, is not based on clinical trials for third line antihypertensive agents. There is general consensus that resistant HTN is due to excessive sodium retention and thus "further diuretic therapy" may be an effective treatment. The choice that one type of diuretic will be superior to another has however not been studied and is usually prescribed in a trial and error manner with diuretics that primarily target the distal nephron (thiazide-like diuretic or spironolactone).

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients aged ≥18 years of age
* Patients will all have hypertension that is not controlled to home target: SBP >135 mmHg and/or DBP >85 mmHg on therapy with one or more antihypertensive drugs for at least 3 months.
* Able to attend one of the three study centres

Exclusion Criteria:

* Inability to give informed consent
* Participation in a clinical study involving an investigational drug or device within 3 months of screening
* Secondary or accelerated hypertension (investigator opinion)
* Diabetes mellitus (Type 1 or type 2)
* eGFR <60 mls/min, hyponatraemia, hypokalaemia
* Pregnancy, breast feeding
* Women of child bearing potential who are unwilling to use effective contraception
* Childbearing potential is defined as women who have experienced menarche and who have not undergone successful surgical sterilisation or who are not post-menopausal (irregular menstrual periods, or amenorrhoea >12 months, with serum follicle stimulating hormone (FSH) >35mIU/ml; women taking hormone replacement therapy (HRT)
* Women of childbearing potential will be eligible if they are willing to use acceptable contraception (combined oral contraceptives, progesterone only contraceptives, intrauterine device, barrier methods) or they are abstinence due to lifestyle choice or their partner is sterile (vasectomy).
* Anticipated change of medical status during the trial (e.g. surgical intervention requiring >2 weeks convalescence)
* Recent (<6 months) cardiovascular event requiring hospitalisation (e.g. myocardial infarction or stroke)
* Requirement for study drug or other loop diuretic for reason other than to treat hypertension
* Clinically relevant contra-indication to treatment with torasemide: hypersensitivity, hereditary problems of glucose intolerance, Lapp lactase deficiency of glucose-galactose malabsorption
* Current therapy for cancer
* Concurrent chronic illness, or other reasons likely to preclude 18-week participation in the study
* Any concomitant condition that, in the opinion of the investigator, may adversely affect the safety and/or efficacy of the study drug or severely limit that patients life-span or ability to complete the study (e.g. alcohol or drug abuse, disabling or terminal illness, severe liver impairment, mental disorders)
* Treatment with any of the following medications -
* Oral corticosteroids within 3 months of screening. Treatment with systemic corticosteroids is also prohibited during study participation
* Chronic stable use, or unstable use of NSAIDs (other than low dose aspirin or occasional OTC analgesic doses) is prohibited. Chronic use is defined as >3 consecutive days of treatment per week. In addition intermittent use of NSAIDs is discouraged throughout the study. For those requiring analgesics during the study, paracetamol or opiate drugs are recommended.
* Use of lithium
* Participants on the following medications may be included provided they meet the following criteria
* Use of thiazide or loop diuretics prior to the study if the diuretic can be stopped for 2 weeks (washout) before the study medication administered.
* The use of short acting nitrates (e.g. sublingual nitroglycerin) is permitted. However, participants should avoid short acting oral nitrates within 4 hours of screening or an subsequent visit
* The use of long acting nitrates (e.g. Isordil) is permitted but the dose must be stable for at least 2 weeks prior to screening and randomisation
* The use of sympathomimetic decongestants is permitted, though not within 24 hours of any study visit/BP assessment
* The use of theophylline is permitted but the dose must be stable for at least 4 weeks prior to screening and throughout the study
* The use of phosphodiesterase type V inhibitors is permitted. However, study participants must refrain from taking these medications for at least 7 days prior to screening or any subsequent study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in ABPM | 16 weeks
  Change in 24h ABPM systolic BP AUC at the end of the 16-week treatment phase compared to baseline

SECONDARY OUTCOMES:
change in 24h ABPM diastolic BP AUC | 16 weeks
  change in 24h ABPM diastolic BP AUC between baseline and the end of treatment
change in day time ABPM systolic and diastolic BP AUC | 16 weeks
  change in day time ABPM systolic and diastolic BP AUC between baseline and the end of treatment
change in night time ABPM systolic and diastolic BP AUC | 16 weeks
  change in night time ABPM systolic and diastolic BP AUC between baseline and the end of treatment
change in HBPM SBP and DBP AUC | 16 weeks
  change in HBPM SBP and DBP AUC over the entire study period
changes in serum electrolytes | 16 weeks
  changes in serum electrolytes over the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Sandosh Padmanabhan, MbChB PhD, Study Chair — University of Glasgow
Locations (1):
- Glasgow Clinical Research Facility, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McCallum L, Lip S, McConnachie A, Brooksbank K, MacIntyre IM, Doney A, Llano A, Aman A, Caparrotta TM, Ingram G, Mackenzie IS, Dominiczak AF, MacDonald TM, Webb DJ, Padmanabhan S. UMOD Genotype-Blinded Trial of Ambulatory Blood Pressure Response to Torasemide. Hypertension. 2024 Oct;81(10):2049-2059. doi: 10.1161/HYPERTENSIONAHA.124.23122. Epub 2024 Jul 30. PMID 39077768
- [Derived] McCallum L, Brooksbank K, McConnachie A, Aman A, Lip S, Dawson J, MacIntyre IM, MacDonald TM, Webb DJ, Padmanabhan S. Rationale and Design of the Genotype-Blinded Trial of Torasemide for the Treatment of Hypertension (BHF UMOD). Am J Hypertens. 2021 Feb 18;34(1):92-99. doi: 10.1093/ajh/hpaa166. PMID 33084880